CLINICAL TRIAL: NCT03166410
Title: Use of Autologous Adipose-Derived Stromal Vascular Fraction To Treat Osteoarthritis of Hip, Knee, Ankle, and Thumb Joints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Plastic Surgery (Industry)
Responsible Party: Principal Investigator, Jaime R. Garza, MD, Principal Investigator, Texas Plastic Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVFOA-01
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Carboxylesterase

ARMS (1):
- Cell Treatment (Experimental)
  Interventions: Procedure: Cell injection

INTERVENTIONS:
Procedure: Cell injection

SUMMARY:
This study will examine the safety and efficacy of autologous adipose-derived stromal vascular fraction (SVF) cells for treatment of hip, knee and thumb osteoarthritis (OA); monitoring adverse events and measuring pain, function and stiffness in the joints of osteoarthritic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Grade II through Grade IV hip, knee, ankle osteoarthritis using Kellgren-Lawrence grading scale (K-L Grade) as diagnosed using weight bearing X-ray, physician review, and/or pre-op MRI
2. Stage II through IV carpometacarpal (CMC) osteoarthritis using Eaton-Little's staging of CMC OA as diagnosed by X-ray and physical examination
3. Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed
4. Subjects with ASA grade I, II, or III
5. Males and females 25-85 years old
6. Subjects must have continued pain in their targeted/treatment joint despite conservative therapies for at least 3 months

Exclusion Criteria:

1. Subjects that are allergic to lidocaine, epinephrine or valium
2. Subjects with a history of bleeding disorders, anticoagulation therapy that cannot be stopped as follows prior to injection; Thrombolytics and anti-platelet medication including but not limited to Coumadin (warfarin) for 3 days, Plavix (clopidogrel) for 3 days, acetylsalicylic acid (ASA)/NSAIDs/fish oil supplements for 7 days, Xeralta® (rivaroxaban) for 24 hours
3. Subjects with systemic immunosuppressant use within six (6) weeks from screening and subjects with HIV/viral hepatitis
4. Subjects with chondrocalcinosis, Paget's disease and Villonodular synovitis
5. Women that are pregnant or planning to become pregnant during the study
6. Subjects on long term use of oral steroids
7. History of any chemotherapy or radiation therapy on the targeted/treatment joint or adipose harvest site

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of Treatment-Emergent Adverse Events | 1 year
  Subjects will be monitored for adverse events

SECONDARY OUTCOMES:
Efficacy - Change in Pain Scores at All Follow-up Visits | 3 months, 6 months, 1 year, 2 years
  Pain scores will be collected at all visits

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Plastic Surgery, San Antonio, Texas, United States